CLINICAL TRIAL: NCT01657045
Title: A Phase I Randomized, Double-Blind, Placebo Controlled Dose Escalation Study to Evaluate the Safety and Efficacy of JVS-100 Administered by Needle-free Dermal Injection to Cohorts of Adults Receiving Surgical Sternotomy Incisions
Brief Title: Study to Evaluate the Safety and Efficacy of Dermal Injections of JVS-100 Given to Adults Receiving Median Sternotomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SironRX Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRX-001
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Median Sternotomy
Keywords: Cicatrix; Wound healing
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Subjects will be randomized to receive injections JVS-100 or placebo.
  Interventions: Biological: JVS-100 or placebo
- Cohort 2 (Experimental): Subjects will be randomized to receive injections JVS-100 or placebo.
  Interventions: Biological: JVS-100 or placebo
- Cohort 3 (Experimental): Subjects will be randomized to receive injections of JVS-100 or placebo.
  Interventions: Biological: JVS-100 or placebo

INTERVENTIONS:
Biological: JVS-100 or placebo — Injections will be delivered depending on sternal incision length.
  Arms: Cohort 1
Biological: JVS-100 or placebo — Injections will be delivered depending on sternal incision length.
  Arms: Cohort 2
Biological: JVS-100 or placebo — Injections will be delivered depending on sternal incision length.
  Arms: Cohort 3

SUMMARY:
This study will investigate the safety and efficacy of using JVS-100 to accelerate wound healing and reduce scar formation in subjects receiving surgical incisions ("sternotomies") during cardiovascular surgery. Twenty-five (25) subjects receiving a median sternotomy of 16 - 25 cm in the process of cardiothoracic surgery will be enrolled consecutively and be followed for 6 months post-dosing. Three cohorts of approximately 8 subjects each will be enrolled, and within each cohort subjects will be randomized 3:1 to receive a single set of needle-free dermal injections of either JVS-100 or placebo. JVS-100 or placebo will be delivered along the edge of the sternal wound using a needle-free injection device that has FDA-clearance for subcutaneous injections.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 40 - 80 years of age inclusive
* Patients undergoing median sternotomy for cardiac surgical procedures, with incision length of 16-25 cm
* Subject must be able to understand the study procedures, agree to participate in the study program, and voluntarily provide written informed consent
* Subjects with BMI 25 - 40 kg/m2
* All subjects age 50 or older must have had a Fecal occult blood test (FOBT) or fecal immunochemical test (FIT) that was negative within the last year or a colonoscopy within the last 10 years
* Women age 40 - 65 must have had a Papanicolaou (PAP) test that was negative within the last 5 years unless a total hysterectomy has been previously performed for benign disease
* Women age 40 or older must have had a mammogram that was negative within the last year
* All diabetic subjects must have had an ophthalmologic exam within the last year showing no active proliferative retinopathy.

Exclusion Criteria:

* Subject is scheduled for mechanical device assistance or, heart transplantation
* Class IV heart failure
* Subject had acute myocardial infarction less than 3 days prior to scheduled surgery
* Subject is undergoing urgent bypass surgical procedure
* History of scleroderma, a connective tissue disorder, rheumatoid arthritis, or ankylosing spondylitis or systemic lupus erythematosus (SLE)
* Pregnant or lactating women or subjects of childbearing potential not protected by an effective method of birth control
* Life expectancy of < 1 year
* Diabetes mellitus with HgbA1C >10.5% tested within 2 weeks prior to surgery
* Existing scarring in the area of study
* Subject has received a cytotoxic agent or has a history of chest radiation therapy and/or will likely require such treatment in the 30 day period following surgery, not including use of radiation for diagnostic imaging, e.g., PET Scan, CT SCAN, Fluro, Myocardial Perfusion (SPECT).
* Chest tattoos over the sternum, breast implants, prior mastectomies or lumpectomies
* Subject plans to use an alternative/accessory wound healing treatment
* Infection being treated with systemic antibiotics within 3 days of scheduled surgery
* Chronic kidney disease (stage 5) requiring dialysis
* Significant Hepatic disease
* Significant is known to be infected with HBV, HIV or HCV
* Clinically significant elevations or decreases in PT/PTT/INR/WBC
* Concurrent medical condition that is associated with prolonged recovery from surgery (e.g., significant respiratory disease, high risk for ventilator dependence, current use of systemic steroids)
* Subject has cognitive impairment
* Any patient with a history of cancer with the exception of: 1) The cancer was limited to curable non-melanoma skin malignancies; 2) The cancer was removed by a successful tumor resection, with or without radiation or chemotherapy treatment, 5 years or more prior to enrollment in this study without recurrence.
* Men unwilling to agree to barrier contraception unless previously received a vasectomy
* Presence of any other condition that, in the opinion of the investigator, might compromise any aspect of the trial
* Previous treatment with an angiogenic growth factor or with stem cell therapy within 1 year
* Participation in another clinical trial of an investigational agent in the previous 30 days
* History of drug or alcohol abuse in the past year

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of ascending doses of JVS-100 delivered via needle-free dermal injections to subjects receiving surgical incisions following cardiothoracic surgery. | 6 months

SECONDARY OUTCOMES:
To investigate the preliminary efficacy of ascending doses JVS-100 delivered via needle-free dermal injections to subjects receiving surgical incisions following cardiothoracic surgery. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amit Patel, MD, Principal Investigator — University of Utah; Robert Michler, MD, Principal Investigator — Montefiore Medical Center
Locations (6):
- United States (6):
  - Pepin Heart Institute, Tampa, Florida
  - Northwestern University Bluhm Cardiovascular Inst, Chicago, Illinois
  - Montefiore Medical Center, New York, New York
  - Summa Health System Hospital, Akron, Ohio
  - University of Utah Hospital, Salt Lake City, Utah
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia